CLINICAL TRIAL: NCT02264054
Title: Investigation of Metabolism and Pharmacokinetics of Talsaclidine After Administration of Single Oral and Single Intravenous Dose of 20 mg of [14C]-Labelled Talsaclidine to 6 Healthy Subjects
Brief Title: Pharmacokinetics of Talsaclidine After Administration to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 506.109
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- [14C]talsaclidine, oral (Experimental): single dose of 20 mg oral solution
  Interventions: Drug: [14C]talsaclidine, oral
- [14C]talsaclidine, iv (Active Comparator): single dose of 20 mg intravenous (iv) infusion
  Interventions: Drug: [14C]talsaclidine, iv

INTERVENTIONS:
Drug: [14C]talsaclidine, oral
  Arms: [14C]talsaclidine, oral
Drug: [14C]talsaclidine, iv
  Arms: [14C]talsaclidine, iv

SUMMARY:
Study to investigate metabolism, pharmacokinetic, safety and tolerability of talsaclidine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age range from 50 to 65 years
* Participants should be within 20% of their normal weight (Broca-Index)
* Written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Results of the medical examination or laboratory tests (especially those which indicate liver malfunction) are judged by the clinical investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Disease of the central nervous system (such as epilepsy) or with psychiatric disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (≥ 24 hours) within one month before enrolment in the study
* Intake of any other drugs which might influence the results of the trial during the week previous the start of the study
* Participation in another study with an investigational drug within the last 2 months preceding this study
* Unability to refrain from smoking on study days
* Volunteers who smoke more than 10 cigarettes (or 3 cigars or pipes) per day
* Volunteers who drink more than 40 g of alcohol per day
* Volunteers who are dependent on drugs
* Blood donation ((≥ 100 ml) within the last 4 weeks
* Excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1999-02; Primary Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
[C14]-radioactivity concentration in blood | up to 96 hours after drug administration
[C14]-radioactivity concentration in plasma | up to 96 hours after drug administration
[C14]-radioactivity concentration in urine | up to 96 hours after drug administration
Area under the plasma concentration-time curve (AUC) | up to 96 hours after drug administration
Terminal half-life (t1/2) | up to 96 hours after drug administration
Maximum concentration of the analyte in plasma (Cmax) | up to 96 hours after drug administration
Time to reach maximum plasma concentration (tmax) | up to 96 hours after drug administration
Absolute bioavailability based on AUC | up to 96 hours after drug administration
Drug absorption (fa) based on radioactivity | up to 96 hours after drug administration

SECONDARY OUTCOMES:
Urinary excretion (Ae) | up to 96 hours after drug administration
Mean residence time (MRT) | up to 96 hours after drug administration
Apparent clearance (CL) | up to 96 hours after drug administration
Apparent volume of distribution (Vz/f)) | up to 96 hours after drug administration
Plasma protein binding of the [14C] radioactivity | up to 96 hours after drug administration
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 8 days after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant findings in electrocardiogram | up to 8 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after last drug administration